CLINICAL TRIAL: NCT06175832
Title: PPOS and CFA for Elective Freeze-all Ovarian Stimulation Cycles: a Prospective Cross-over Study
Brief Title: PPOS (Progestin Primed Ovarian Stimulation) and Corifollitropin Alfa (CFA) Cross-over Study
Acronym: P-CCROSS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ONZ-2023-0299; 2023-506694-35-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-28; First posted 2023-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Stimulation; Quality of Life; Preimplantation Genetic Testing; Fertility Preservation
MeSH Terms: interventions — follitropin beta; ganirelix; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CFA/PPOS cycle (Experimental): Interventional stimulation
  Interventions: Drug: Elonva®; Drug: Puregon®; Drug: Gonapeptyl®; Drug: Cerazette®
- rFSH / GnRH antagonist cycle (Active Comparator): Conventional stimulation
  Interventions: Drug: Puregon®; Drug: Orgalutran®; Drug: Gonapeptyl®

INTERVENTIONS:
Drug: Elonva® — Single injection
  Arms: CFA/PPOS cycle
Drug: Puregon® — Multiple injections
Drug: Orgalutran® — Multiple injections
  Arms: rFSH / GnRH antagonist cycle
Drug: Gonapeptyl® — Double injection
Drug: Cerazette® — Oral tablet
  Arms: CFA/PPOS cycle

SUMMARY:
P-CCROSS is a randomized, prospective monocentric phase 4 study with a crossover study design. The aim of the study is to compare patient satisfaction (by means of questionnaires) and treatment compliance with IVF treatment with CFA (corifollitropin alfa) and PPOS (Progestin-Primed Ovarian Stimulation) versus conventional IVF treatment with a recombinant FSH/GnRH antagonist. The study will also compare patients undergoing elective fertility preservation versus PGT-A (pre-implantation genetic testing for aneuploidy) patients.The study will have a crossover design so that patients will receive both forms of treatment. The investigators will also compare the endocrine profile and ovarian response of CFA/PPOS versus rFSH/GnRH ovarian stimulation cycles.

ELIGIBILITY:
Prescreening: Clarification: Pre-screening might be performed to identify women with AFC > 5 and AMH > 1.1 ng/ml (Bologna criteria, AFC and AMH values are valid for one year).

Inclusion criteria for:

* Group 1: indication for oocyte cryopreservation
* Group 2: indication for IVF/ICSI and PGT-A

Inclusion criteria for both groups:

* First ovarian stimulation cycle
* Aged ≥ 18 and < 41 years old at the time of first OPU

Exclusion Criteria:

* contra-indication for ovarian stimulation
* expected poor ovarian response (Bologna Criteria)
* PCOS patients
* refusal to fill out questionnaires before, during and after treatment
* simultaneous participation in another clinical study
* untreated and uncontrolled thyroid dysfunction;
* current use of oral contraceptives, anti-psychotics, anti-epileptics or chemotherapy;
* pregnant or breastfeeding women. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related quality of life and patient satisfaction after comparing two different ovulation stimulation cycles | Six months
  Comparison of CFA / PPOS stimulation versus conventional rFSH / GnRH antagonist ovarian stimulation cycles with respect to mean treatment-related quality of life and patient satisfaction. Treatment-related quality of life and patient satisfaction retrieved from the second questionnaire (Q2), which is completed at the end of each stimulation cycle; after the agonist trigger and before the oocyte retrieval.Q2 is a combination of the treatment module of the validated FertiQoL questionnaire and the EFESO questionnaire. This questionnaire will assess the environment and tolerability of the fertility treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No